CLINICAL TRIAL: NCT05180773
Title: Randomized Evaluation of Bromocriptine In Myocardial Recovery THerapy for Peripartum Cardiomyopathy (REBIRTH)
Brief Title: Impact of Bromocriptine on Clinical Outcomes for Peripartum Cardiomyopathy
Acronym: REBIRTH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dennis M. McNamara, MD, MS (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Dennis M. McNamara, MD, MS, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY21090058; UG3HL153847 (NIH)
Record Dates: First submitted 2021-12-09; First posted 2022-01-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-02

CONDITIONS: Peripartum Cardiomyopathy, Postpartum
MeSH Terms: conditions — Peripartum Cardiomyopathy | interventions — Bromocriptine; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: 200 women meeting all inclusion and exclusion criterial will be randomized in a placebo controlled double blind investigation evaluating the impact of bromocriptine on outcomes for women newly diagnosed with peripartum cardiomyopathy. An additional 50 women in excluded from the trial due to an intent to continue breastfeeding but meeting all other criteria will be enrolled in an observational cohort. All women with receive standard medical care for peripartum cardiomyopathy and will be followed for up to three years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Once consent is obtained the screening sheet will be submitted to the data coordinating center. This will be reviewed to ensure the subject meets criteria for randomization. Subjects will be randomized by the Data Coordinating Center (DCC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bromocriptine Treatment Arm (Active Comparator): 100 Women in the Treatment Arm will receive guideline directed medical therapy for heart failure plus 8 weeks of bromocriptine administered orally as 2.5 mg twice daily for 2 weeks then 2.5mg once daily for 6 weeks. Women not on clinical anticoagulation will also receive prophylactic anticoagulation with rivaroxaban 10 mg once daily for 8 weeks while on bromocriptine.
  Interventions: Drug: Bromocriptine; Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT); Drug: Rivaroxaban
- Placebo Arm (Placebo Comparator): 100 Women in the Placebo Arm will receive guideline directed medical therapy for heart failure plus 8 weeks of a placebo administered orally twice daily for 2 weeks then once daily for 6 weeks. Women not on clinical anticoagulation will not receive rivaroxaban but will instead receive a second placebo for 8 weeks.
  Interventions: Drug: Placebo; Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT); Drug: Second Placebo
- Breastfeeding Observational Cohort (Other): Up to 50 women meeting all other criteria but excluded from REBIRTH due to an intent to continue to breastfeed will be enrolled in an observational cohort. They will receive guideline directed medical therapy with no additional interventions and will have the same follow up and assessment of myocardial recovery by echocardiogram at 6 and 12 months post entry as women in the randomized trial.
  Interventions: Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT)

INTERVENTIONS:
Drug: Bromocriptine — Bromocriptine 2.5 mg one tablet by mouth twice daily for 2 weeks then once daily for 6 weeks. Subjects not on anticoagulation at the time of entry will also receive rivaroxaban 10 mg tablets once daily for 8 weeks while on bromocriptine.
  Other Names: Parlodel; Cycloset
  Arms: Bromocriptine Treatment Arm
Drug: Placebo — Placebo one tablet by mouth twice daily for 2 weeks then once daily for 6 weeks. Subjects who are not on anticoagulation will not receive rivaroxaban but will receive a second placebo once daily for 8 weeks while on study drug.
  Arms: Placebo Arm
Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT) — GDMT will potentially include angiotensin converting enzyme inhibitors (ACEi), angiotensin II receptor antagonists (ARB), angiotensin receptor blocker-neprilysin inhibitors (ARNI), beta adrenergic receptor antagonists (beta blockers) , Mineralocorticoid receptor antagonists (MRA), sodium-glucose cotransporter-2 inhibitors (SGLT2i),
Drug: Rivaroxaban — Subjects not on anticoagulation clinically who are randomized to bromocriptine will receive rivaroxaban 10 mg tablets once tablet by mouth daily for 8 weeks while on bromocriptine.
  Other Names: Xarelto
  Arms: Bromocriptine Treatment Arm
Drug: Second Placebo — Subjects not on anticoagulation clinically who are randomized to placebo (rather than bromocriptine) will receive a second placebo one tablet by mouth daily for 8 weeks.
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
The study will enroll 200 women newly diagnosed with peripartum cardiomyopathy within 5 months postpartum in a randomized placebo controlled trial of bromocriptine therapy to evaluate its impact on myocardial recovery and clinical outcomes. Given that bromocriptine prevents breastfeeding, an additional 50 women with peripartum cardiomyopathy excluded from the trial due to a desire to continue breastfeeding but meeting all other entry criteria will be followed in an observational cohort.

DETAILED DESCRIPTION:
The study will enroll 200 women newly diagnosed with peripartum cardiomyopathy within 5 months postpartum in a randomized trial of bromocriptine therapy to evaluate its impact on myocardial recovery. All women will have an assessment of LVEF demonstrating an LVEF < or = 0.40 within 4 weeks prior to consent. The women in the breastfeeding cohort will have a qualifying LVEF < 0.40 within 8 weeks prior to consent. At entry they will then have an assessment of LVEF by echocardiogram which will be repeated at 6- and 12-months post study entry. Subjects in the randomized trial will be randomized to standard medical therapy for heart failure plus placebo or standard therapy plus 8 weeks of bromocriptine (2.5 mg twice daily for 2 weeks then once 2.5 mg daily for 6 weeks). Women receiving bromocriptine not currently on anticoagulation will also receive prophylactic anticoagulation with rivaroxaban 10 mg once daily for 8 weeks.

Primary analysis will compare LVEF at 6 months post entry in the women receiving standard therapy plus bromocriptine to those on standard therapy plus placebo (controlling for initial baseline LVEF). Secondary endpoints will analyze the LVEF in both treatment groups at 12 months post randomization. In addition, subjects will be followed for up to 3 years post randomization and survival free from a major event (cardiac transplantation or durable LVAD implantation) and survival free from heart failure hospitalization will be compared by treatment group.

The benefits of bromocriptine are theoretically related to suppression of prolactin secretion. Breastfeeding increases prolactin levels, and whether continued breastfeeding will impact myocardial recovery in women with peripartum cardiomyopathy remains unknown. As bromocriptine prevents breastfeeding, women who want to continue breastfeeding are excluded from the randomized trial. Up to 50 women meeting all other criteria but excluded from REBIRTH due to an intent to continue to breastfeed will be enrolled in an observational cohort. They will receive standard therapy with no additional intervention and will have the same follow up and assessment of myocardial recovery by echocardiogram at 6- and 12-months post entry as women in the randomized trial.

Blood will be obtained at entry for DNA banking, and analysis of serum, and whole blood RNA . Additional serum and whole blood RNA will be banked at 1-, 3-, and 6-months post randomization. This investigation will evaluate the impact of bromocriptine therapy on the levels of intact 23 kilodalton (kDa) prolactin and the 16 kDa prolactin fragment, as well as microRNA (miR) 146a. The biomarker analysis will also be performed in the observational cohort of women excluded due to continued breast feeding. The impact of these biomarkers on outcomes in both the treatment and control groups as well as the observational cohort excluded due to breastfeeding will be examined.

A core laboratory will analyze all echocardiograms. In addition to quantifying the LVEF at entry, 6 months and 12 months post entry, the core will evaluate global longitudinal strain (LGS) and remodeling (LV volumes) at entry as predictors of outcome and drug response. They will also evaluate the impact of therapy on LGS and LV volumes at 6- and 12-months post randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Presentation with a new diagnosis of peripartum cardiomyopathy
2. Post-delivery and within the first 5 months post-partum.
3. Clinical assessment of an LVEF < or =0.40 within 4 weeks of consent for randomized control trial
4. Clinical assessment of an LVEF < or =0.40 within 8 weeks of consent for breastfeeding cohort
5. Age > or = 18.

Exclusion Criteria:

1. Previous diagnosis of cardiomyopathy, valvular disease or congenital heart disease (with the exception of women with a history of peripartum cardiomyopathy with complete recovery and a documented LVEF > 0.55 prior to or in early pregnancy)
2. Refractory hypertension (Systolic >160 or Diastolic > 95) either at the time of enrollment or at the time of the qualifying LVEF.
3. Postpartum women currently breastfeeding and planning to continue.
4. Evidence of coronary artery disease (>50% stenosis of major epicardial vessel or positive non-invasive stress test)
5. Previous cardiac transplant
6. Current durable LVAD support
7. Currently requiring support with extracorporeal membrane oxygenation (ECMO)
8. Current history of alcohol or drug abuse
9. Chemotherapy or chest radiation within 5 years of enrollment
10. Evidence of ongoing bacterial septicemia
11. Medical, social or psychiatric condition which limit the ability to comply with follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women recently diagnosed with peripartum cardiomyopathy who are 18 years or older and are within 5 months of postpartum.
Enrollment: 250 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) at 6 months post entry as determined by echocardiography | 6 months

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) at 12 months post entry as determined by echocardiography | 12 months
Survival free from cardiac transplantation or implantation of a durable left ventricular assist device (LVAD) | 3 years
Survival free from heart failure hospitalization | 3 years

OTHER OUTCOMES:
Global longitudinal strain (GLS) at 6 months post entry as determined by echocardiography | 6 months
Global longitudinal strain (GLS) at 12 months post entry as determined by echocardiography | 12 months
Left ventricular volumes at 6 months post entry as determined by echocardiography | 6 months
Left ventricular volumes at 12 months post entry as determined by echocardiography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis McNamara, Principal Investigator — University of Pittsburgh
Locations (64):
- United States (64):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine Health, Orange, California
  - Stanford University, Stanford, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois Health Heart Center, Chicago, Illinois
  - Indiana University/Indiana University Health, Indianapolis, Indiana
  - Ascension St. Vincent Heart Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - University of Kentucky, Gill Heart & Vascular Institute, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Karen L Florio, MD, Columbia, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Albert Einstein College of Medicine/ Montefiore Medical Center, The Bronx, New York
  - Atrium Health Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma university Health Science Center, Oklahoma City, Oklahoma
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple Heart and Vascular Institute, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Vanderbilt, Nashville, Tennessee
  - UT Southern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health San Antonio, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Inova Healthcare Services, Fairfax, Virginia
  - Old Dominion University, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Madison, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Quesada O, Scantlebury DC, Briller JE, Michos ED, Aggarwal NR. Markers of Cardiovascular Risk Associated with Pregnancy. Curr Cardiol Rep. 2023 Feb;25(2):77-87. doi: 10.1007/s11886-022-01830-1. Epub 2023 Feb 6. PMID 36745273
- [Derived] Briller JE. Echocardiographic Screening in Hypertensive Pregnancy Disorders: Probing the Window of Opportunity. J Am Coll Cardiol. 2022 Oct 11;80(15):1477-1479. doi: 10.1016/j.jacc.2022.08.717. No abstract available. PMID 36202537

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT05180773/SAP_000.pdf